CLINICAL TRIAL: NCT04813744
Title: Investigation of Atraumatic Restorative Treatment by in Vivo and in Vitro Methods in Terms of the Microbiological, Marginal Adaptation and Microleakage
Brief Title: Microbiological and Microscopic Evaluation of Atraumatic Restorative Treatment in Adult Dentition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Tekbas Atay, Project manager, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1432
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Dentin Caries; Infection
Keywords: Atraumatic restorative treatment; Glass ionomer cement; Marginal adaptation
MeSH Terms: conditions — Infections | interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Intervention Model Description: The clinical studies were carried out in the occlusal dentin caries of 25 permanent molar teeth in participants with high caries risk and between 19-35 years of age. The caries tissue were removed with hand instruments in accordance procedure of atraumatic restorative treatment. Then the total counts of bacteria, facultative anaerobe bacteria, Mutans Streptococci, and Lactobacilli supp. counts in the affected dentin were evaluated quantitatively. The weights of samples were measured with an electronic balance (Shimadzu, Type AX200, Japan). The cavities were restored with a glass ionomer cement (KetacTM Molar Easymix, ESPE Dental AG, Seefeld, Germany). Twenty replicas of randomly selected ART restorations were prepared and marginal adaptation was evaluated by scanning electron microscopy. After 6 months, the same protocols were repeated. Data were analyzed with Paired Sample and Wilcoxon Paired t-tests, Pearson, Spearman correlation, and Chi-Square tests (p< 0.05).
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigation of atraumatic restorative treatment in adults with a high risk of caries (Experimental): The study group included a total of 25 healthy individuals with high caries risk who had molar teeth in their mouth with 3-4 mm depth occlusal dentin caries. In the clinical study, the infected and demineralized dentin was cleaned manually with a sterile excavator. The dentin sample was taken from the last removable and affected dentin layer at the cavity floor by one excavation for microbiological assessment. The teeth were restored with a conventional glass ionomer cement. In the 6th month, restorations were removed by using low-speed round steel bur, and the dentin samples were removed with an excavator from the cavity floor to repeat the microbiological assessment. In the first week and 6th month of atraumatic restorative treatment, the impressions were taken from the restored teeth to prepare replicas. The replicas of the twenty teeth out of 25 were randomly selected to evaluate of marginal adaptation under scanning electron microscopy.
  Interventions: Procedure: Atraumatic restorative treatment

INTERVENTIONS:
Procedure: Atraumatic restorative treatment

SUMMARY:
Atraumatic Restorative Treatment (ART) was proposed as a new and effective method in the 1990s to provide conservative dental treatment to the people living in economically underdeveloped countries, due to lack of dental treatment facilities. In the technique, after the carious dentin is removed by excavation with hand instruments, the powder-liquid system conventional glass ionomer cement (GIC) which does not require special devices for mixing and hardening is used as a filling material. Because of these advantages of the treatment, the usage fields of ART have been expanded considering that it can be applied in the cases that working with rotary instruments is difficult or even impossible. But only a few research has been conducted on ART in adults and it must be investigated in terms of the clinical safety of ART by the studies focused on the counts and activities of the microorganisms in carious dentin left on the cavity floor. The purpose of this study is to investigate the reliability of ART in adult individuals related to the marginal adaptation of the restorations and the microbiological changes in the left carious dentin using in vitro and in vivo methods. In the in vivo part of the study, occlusal dentin carious of 25 participants at high risk of caries were removed with hand instruments and microorganisms of the last removed carious dentin were evaluated quantitatively concerning the bacterias playing a major role in caries lesions. The restorations of the teeth were carried out using ART technique with a GIC which has been proven its effectiveness in preventing the caries progression and recurrent caries in the practice of dentistry for many years. After six months, the microbiological assessment was repeated such as baseline. Marginal adaptation and the presence of the gaps in the ART restorations on the replicas created with the impression materials at the baseline and sixth month were investigated under scanning electron microscope. At the end of the study, the teeth were restored by the conventional methods and using composite material.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* 19-35 years of age;
* Good general health;
* High risk of caries;
* No evident signs of occlusal parafunctions.

Tooth:

* Molar tooth;
* 3-4 mm depth occlusal dentin caries;
* Vital;
* In occlusion;
* Proper tooth axes.

Exclusion Criteria:

Patient:

* Using regular medication;
* Pregnancy or lactation;
* Received radiotherapy or chemotherapy;
* Tooth clenching, bruxism.

Tooth:

* Spontaneous pain;
* Radiographic alterations in the periapical region;
* Presence of tooth mobility;
* Previously restored;
* Broken and/ or cracked.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-05-09 (Actual); Primary Completion 2011-03-03 (Actual); Study Completion 2011-03-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of microbiological parameters | 6 months
  Change at the counts of microorganisms
Microscopic analyses of the marginal gap formation | 6 months
  Change at the marginal integrity of restorations

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Tekbas Atay, PhD, Principal Investigator — Department of Restorative Dentistry, Faculty of Dentistry, Trakya University, Edirne, Turkey; Fatma Koray, Prof. Dr., Study Chair — Department of Restorative Dentistry, Faculty of Dentistry, Yeniyüzyıl University, Istanbul, Turkey

IPD SHARING:
Plan to Share IPD: No